CLINICAL TRIAL: NCT05794737
Title: Immunohistochemical Expression of Inhibin Beta A (INHBA) in Colorectal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mera Atef Fayez, Teaching Assistant of Pathology, Sohag University
Other Study IDs: Soh-Med-23-03-08MS
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
Keywords: Inhibin Beta A; Colorectal Carcinoma; Immunohistochemistry
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 60 formalin fixed, Paraffin embedded Colorectal Cancer tissue blocks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: 60 archived Formalin-fixed Paraffin-embedded tissue blocks of Colorectal Carcinoma will be obtained and sectioned. From each block; Two tissue sections will be prepared, one tissue section will be stained by Hematoxylin and Eosin to detect tumor phenotype and depth of invasion. Other tissue section will be immunohistochemically stained by Anti-Human INHBA.
  Interventions: Biological: Immunohistochemical staining

INTERVENTIONS:
Biological: Immunohistochemical staining — Staining of Colorectal Carcinoma tissue sections by monoclonal antibodies against human Inhibin Beta A by immunohistochemical procedures.

SUMMARY:
A retrospective observational study to evaluate immunohistochemical expression of Inhibin Beta A (INHBA) in 60 cases of Colorectal Carcinoma, and compare levels of its expression to different clinicopathological criteria.

DETAILED DESCRIPTION:
Colorectal Carcinoma is an aggressive malignant epithelial tumor with an observable high incidence. Tumor invasion and metastasis to distant sites are two important issues which determine patient's outcome, so detecting novel biological markers that are involved in tumor proliferation and invasion with subsequent targeting by future medical drugs will positively improve patient's prognosis.

Inhibin Beta A (INHBA) is a glycoprotein molecule that has a role in tumor cells proliferation and invasion in different human malignancies. The aim of this study is to detect expression of INHBA in 60 archived formalin-fixed Paraffin-embedded tissue blocks of patients suffered from Colorectal Carcinoma, and to correlate different levels of its expression to some studied clinical and pathological criteria (Age, Sex, Tumor size, location, depth of tumor invasion, status of regional lymph nodes, vascular and perineural invasion).

ELIGIBILITY:
Inclusion Criteria:

Specimens from patients with Colorectal Carcinoma. Tissue blocks with sufficient material. Specimens with sufficient clinical data.

Exclusion Criteria:

Tissue blocks with insufficient, destroyed or necrotic material. Specimens with insufficient clinical data.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Archived Formalin-fixed, Paraffin-embedded tissue blocks belonged to patients suffered from colonic and/or rectal cancers. Patients were admitted to sohag university hospital and underwent colectomy and their colonic specimens were sent to Pathology Laboratory of the same hospital to ascertain diagnosis and tumor phenotype, from period Janurary 2021 to December 2022.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Detection of INHBA in Colorectal Carcinoma. | 6 months
  Detection of expression of INHBA in Colorectal Carcinoma cells by immunohistochemical approach, using anti-human INHBA monoclonal antibody.

SECONDARY OUTCOMES:
Correlation between INHBA expression in Colorectal Carcinoma and clinicopathological parameters. | 6 months
  Correlation between different levels of INHBA expression in Colorectal Carcinoma cells and some clinical and pathological parameters as age, sex, tumor phenotype and nodal status.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided